CLINICAL TRIAL: NCT01329783
Title: Incidence And Risk Factors For Acquired Immune Deficiency Syndrome (AIDS) Defining And Non-AIDS Defining Malignancies, And Other AIDS Defining Illnesses In The EuroSIDA Study
Brief Title: EuroSIDA As An External Comparator To MOTIVATE Trials
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: Copenhagen HIV Programme (Other Government); Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A4001104
Record Dates: First submitted 2011-03-16; First posted 2011-04-06 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EuroSIDA sub-cohort: HIV infected patients in the EuroSIDA cohort who meet the entry criteria for maraviroc pivotal clinical trials (MOTIVATE 1 and MOTIVATE 2)
  Interventions: Other: maraviroc

INTERVENTIONS:
Other: maraviroc — No intervention is distributed during this trial.
  Other Names: Selzentry, Celsentri

SUMMARY:
Human Immunodeficiency Virus (HIV) infected patients who meet the entry criteria for the maraviroc pivotal trials (Maraviroc versus Optimized Therapy in Viremic Antiretroviral Treatment-Experienced Patients, MOTIVATE) will be identified from the EuroSIDA HIV cohort. The rates of specific clinical adverse events in this identified patient population will be compared with the rates of these events in the participants of the MOTIVATE trials.

DETAILED DESCRIPTION:
All patients in EuroSIDA cohort that meet the entry criteria of MOTIVATE trials are included without any sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 16 at baseline.
* Viral Load (VL) > 5000 copies/ml at baseline (and measured in 6 months prior to baseline).
* No changes in antiretroviral (ARV) regimens in the month period prior to baseline, or on no ARVs in the month prior to baseline.
* > 3 months exposure (sequential or cumulative) to at least 3 of the following;
* Any nucleoside or nucleotide reverse transcriptase inhibitor (NRTI)
* Non-nucleoside reverse transcriptase inhibitor (NNNRTI)
* Protease Inhibitor (PI )
* Enfuvirtide

Exclusion Criteria:

None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patient aged over 16 at baseline.
  * Viral Load (VL) > 5000 copies/ml at baseline (and measured in 6 months prior to baseline).
  * No changes in antiretroviral (ARV) regimens in the month period prior to baseline, or on no ARVs in the month prior to baseline.
  * > 3 months exposure (sequential or cumulative) to at least 3 of the following;
  * Any nucleoside or nucleotide reverse transcriptase inhibitor (NRTI)
  * Non-nucleoside reverse transcriptase inhibitor (NNNRTI)
  * Protease Inhibitor (PI )
  * Enfuvirtide
Sampling Method: Non-Probability Sample
Enrollment: 1181 (Actual)
Dates: Start 2007-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Malignancy | Median follow up of 3 years
Opportunistic infection | Median follow up of 3 years
Myocardial infarction | Median follow up of 3 years
All cause death | Median follow up of 3 years
Liver related death | Median follow up of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001104&StudyName=EuroSIDA%20As%20An%20External%20Comparator%20To%20MOTIVATE%20Trials